CLINICAL TRIAL: NCT03688438
Title: Post Operative Wound Complications in Patients With BMI ≥35kg/m2 After Posterior Lumbar Spine Surgery: a Randomized Clinical Trial of Closed-Incision Negative-Pressure Therapy
Brief Title: WoundVac in Obese Patients Undergoing Lumbar Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Norton Leatherman Spine Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18.1023
Record Dates: First submitted 2018-09-26; First posted 2018-09-28 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Obesity; Lumbar Spine Surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: Two study arms: (1) Standard of Care and (2) WoundVac
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard of Care (No Intervention): Standard of care wound closure and dressing No active interventions
- WoundVAC (CINPT) (Experimental): Closed-Incision Negative-Pressure Therapy
  Interventions: Device: Closed-Incision Negative-Pressure Therapy

INTERVENTIONS:
Device: Closed-Incision Negative-Pressure Therapy — A foam or gauze dressing is put directly on the wound. This foam acts as a filter to keep any large particles (such as blood clots or dead, sloughed off tissue) from clogging the vacuum system. A clear, occlusive, adhesive film covers and seals the dressing and wound, creating an airtight seal. A drainage tube leads from under the adhesive film and connects to a portable vacuum pump. This pump removes air pressure over the wound. The pump is programmed for strength of suction, amount of time it is to be applied and if it is to be intermittent or continuous. A chamber on the pump collects drainage and moisture is drawn away from the wound site.
  Other Names: WoundVac
  Arms: WoundVAC (CINPT)

SUMMARY:
This is an open label, randomized clinical trial of Closed-Incision Negative-Pressure Therapy to decrease post-operative wound complications in patients with BMI ≥35kg/m2 after posterior lumbar spine surgery.

DETAILED DESCRIPTION:
Methods:

Study Design: Prospective open-label randomized clinical trial of CINPT in obese patients. Subjects will be randomized in a 1:1 to Standard of Care (SOC) and CINPT.

Study Arms: (1) Standard of Care (2) CINPT Sample Size: Based on 30% incidence of wound complications in obese patients undergoing lumbar spine surgery, a sample size of 124 (62 in each cohort) will be needed to detect a decreased incidence of 10% with an α of 0.05 and β of 0.2.

Randomization: Randomization will be done with varying blocks of 4, 6 and 8 using opaque sealed envelopes.

Procedures: All patients will receive standard pre operative prophylactic antibiotics with 2g - 3g Cefazolin or 1g Clindamycin (if patient has known penicillin allergy) based on weight 60 min before incision is made. They will be clipped if needed before being prepped. Each patient will be prepped with alcohol and then either duraprep, chloraprep, or betadine. After the procedure is complete, a subfascial and subcutaneous closed suction drain will be placed in the wound prior to closure. 1 to 3 gram of Vancomycin powder will be placed in the wound. The wound is closed with #1vicryl for the fascial layer followed by 2-0 Vicryl for the subcutaneous layer followed by 3-0 or 4-0 monocryl. In the SOC group, skin glue, Steri-strips, sterile gauze and Tegaderm will be applied to the wound. In the CINPT group, a CINPT dressing will be placed and attached to a compact portable negative pressure unit to deliver 125mmHg continuous pressure for 5 to 7 days. All patients will receive standard wound care instructions before hospital discharge. Patients will return to the clinic in 6±1 days for a wound check and removal of the CINPT.

Primary endpoint: The primary endpoint is the occurrence of a wound complication. A wound complication can include a local inflammatory reaction, wound dehiscence, skin blistering/necrosis, stitch abscess or Incision and drainage for hematoma seroma, deep or superficial infection

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged ≥18 years old
* Patients undergoing posterior lumbar fusion with or without interbody fusion
* Body Mass Index of ≥35kg/m2
* Able to provide Informed Consent
* No prior lumbar spine surgery

Exclusion Criteria:

* Presence of skin infection or any systemic infection
* Known allergy or sensitivity to silver or acrylic adhesive
* Fragile peri-incisional skin
* Patients on anti-coagulation and/or platelet aggregation inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2018-10-15 (Estimated); Primary Completion 2019-10-15 (Estimated); Study Completion 2020-10-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of wound complication | Within one month after surgery
  A wound complication can include a local inflammatory reaction, wound dehiscence, skin blistering/necrosis, stitch abscess or Incision and drainage for hematoma seroma, deep or superficial infection

SECONDARY OUTCOMES:
Days to dry wound | One month after surgery
  Number of days after surgery it took to have the wound become dry

CONTACTS AND LOCATIONS:
Overall Officials: Charles II H Crawford, MD, Principal Investigator — Norton Leatherman S[ine Center
Locations (1):
- Norton Leatherman Spine Center, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No